CLINICAL TRIAL: NCT04779749
Title: Pregnancy Outcomes According to the Gestational Age of Acquiring COVID-19 : an International Case-control Study
Brief Title: Pregnancy Outcomes According to the Gestational Age of Acquiring COVID-19
Status: Completed | Type: Observational
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Jani Jacques, Head of Gynecology-Obstetrics Department, Brugmann University Hospital
Other Study IDs: PregOutCOV
Record Dates: First submitted 2021-03-01; First posted 2021-03-03 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- COVID positive <20 weeks: Case groups 1 will include pregnant patients infected by SARS-CoV2 before 20 weeks' gestation during the period starting on February 1st 2020 and ending on November 30th 2020.
  Interventions: Other: Data extraction from medical files
- COVID positive >20 weeks: Case groups 2 will include pregnant patients infected by SARS-CoV2 after 20 weeks' gestation during the period starting on February 1st 2020 and ending on November 30th 2020.
  Interventions: Other: Data extraction from medical files
- Control: Patients not infected by SARS-CoV2 during pregnancy during the period starting on February 1st 2020 and ending on November 30th 2020
  Interventions: Other: Data extraction from medical files

INTERVENTIONS:
Other: Data extraction from medical files — Data extraction from medical files

SUMMARY:
A new coronavirus, called severe acute respiratory syndrome coronavirus 2 (SARS-CoV2) appeared in Wuhan, China and it arrived to Europe 2-3 months later. It infected millions of persons and led to the death of thousands until May 2020 where numbers of infections per week decreased significantly. However, starting September, number of infections started to escalate again and continued to rise until now.

Hundreds of good quality articles were published during this period to study the relationship and effects of this virus on pregnancy and vice versa, as well as to determine the adverse neonatal and obstetrical outcomes following the infection. In a case-control study using propensity score matching at the level of age, body mass index and comorbidities (diabetes, hypertension, asthma), pregnant women over 20 week's gestation had significantly higher risk for intensive care unit stay, endotracheal intubation, hospitalization for disease related symptoms and need for oxygen therapy. A new systematic review also demonstrated increased risk for ICU admission in pregnant women compared to non-pregnant women and to non-infected pregnant women.

On the other hand, many researchers have demonstrated that the rates of preterm delivery and cesarean delivery have increased as well, others reported a close relation between SARS-CoV2 infection and preeclampsia or preeclampsia like condition. Enormous effort was done in order to understand adverse outcomes related to this infection, however, most studies included patients in the third or late second trimester. Few studies stratified adverse outcomes of the patients according to the trimester of infection.

ELIGIBILITY:
Inclusion Criteria:

Pregnant women with viable fetus after 10 weeks' gestation and known pregnancy outcome during the period starting on February 1st 2020 and ending on November 30th 2020.

Exclusion Criteria:

All ongoing pregnancies, those with unknown outcomes, those terminated medically or voluntary, as well as patients with spontaneous abortion before the 11th gestational week.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will include all pregnant women with viable fetus after 10 weeks' gestation and known pregnancy outcome during the period starting on February 1st 2020 and ending on November 30th 2020.
Sampling Method: Non-Probability Sample
Enrollment: 10925 (Actual)
Dates: Start 2020-12-08 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Preterm delivery | 5 minutes
  Delivery at a gestational age < 37 weeks
Preeclampsia | 5 minutes
  Preeclampsia is defined as elevated blood pressure (Systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg on at least 2 occasions at least 4 hours apart after 20 weeks of gestation in a previously normotensive patient) and the new onset of 1 or more of the following:
  * Proteinuria ≥0.3 g in a 24-hour urine specimen or protein/creatinine ratio ≥0.3 (mg/mg) (30 mg/mmol) in a random urine specimen or dipstick ≥2+ if a quantitative measurement is unavailable
  * Platelet count <100,000/microL
  * Serum creatinine >1.1 mg/dL (97.2 micromol/L) or doubling of the creatinine concentration in the absence of other renal disease
  * Liver transaminases at least twice the upper limit of the normal concentrations for the local laboratory
  * Pulmonary edema
  * New-onset and persistent headache not accounted for by alternative diagnoses and not responding to usual doses of analgesics
  * Visual symptoms (eg, blurred vision, flashing lights or sparks, scotomata)
Eclampsia | 5 minutes
  Eclampsia is defined by the occurrence of a grand mal seizure in a woman with preeclampsia in the absence of other neurologic conditions that could cause seizure.
Hemolysis Elevated Liver enzymes Low Platelets Syndrome (HELLP) | 5 minutes
  HELLP syndrome is considered to be a serious complication or variant of preeclampsia in pregnant women.
Number of participants with Cesarean delivery (CD) | 5 minutes
  Number of participants with Cesarean delivery (CD)
Percentage of participants with Cesarean delivery (CD) | 5 minutes
  Percentage of participants with Cesarean delivery (CD)
Deep venous thrombosis | 5 minutes
  diagnosed by imaging tools such as venous Doppler ultrasound of the lower limbs
Pulmonary embolism | 5 minutes
  diagnosed by imaging tools such as angio-CT scan of the thorax.
Pregnancy loss at less than 24 weeks' gestation | 5 minutes
Intrauterine Fetal Demise (IUFD) | 5 minutes
  Pregnancy loss at 24 weeks or more, or the delivery of a neonate weighing more than 500 g
Maternal death | 5 minutes
  Maternal death
Low birth weight | 5 minutes
  birth weight at less than 2500g
Number of participants with Neonatal intensive care unit (NICU) admission | 5 minutes
  Number of participants with Neonatal intensive care unit (NICU) admission
Percentage of participants with Neonatal intensive care unit (NICU) admission | 5 minutes
  Percentage of participants with Neonatal intensive care unit (NICU) admission
Number of participants with APGAR score (Activity, Pulse, Grimace, Appearance, Respiration score) at 5 minutes < 7: | 5 minutes
  The score minimum is 0 and maximum is 10. Higher score means better outcome.
Percentage of participants with APGAR score (Activity, Pulse, Grimace, Appearance, Respiration score) at 5 minutes < 7: | 5 minutes
  The score minimum is 0 and maximum is 10. Higher score means better outcome.
Number of participants with Respiratory distress at birth | 5 minutes
  Number of participants with Respiratory distress at birth
Percentage of participants with Respiratory distress at birth | 5 minutes
  Percentage of participants with Respiratory distress at birth
Neonatal death | 5 minutes

SECONDARY OUTCOMES:
Number of participants with Delivery < 32 weeks | 5 minutes
Percentage of participants with Delivery < 32 weeks | 5 minutes
Number of participants with Spontaneous delivery < 37 weeks | 5 minutes
Percentage of participants with Spontaneous delivery < 37 weeks | 5 minutes
Number of participants with Fetal distress | 5 minutes
  referred to bradycardia, recurrent late or variable deceleration on antepartum or intrapartum cardiotocogram.
Percentage of participants with Fetal distress | 5 minutes
  referred to bradycardia, recurrent late or variable deceleration on antepartum or intrapartum cardiotocogram.
Number of participants with Unscheduled cesarean delivery | 5 minutes
Percentage of participants with Unscheduled cesarean delivery | 5 minutes
Postpartum hemorrhage | 5 minutes
  defined as the estimated blood loss of > 500 mL
Number of participants with Intraventricular hemorrhage | 5 minutes
Percentage of participants with Intraventricular hemorrhage | 5 minutes
Umbilical cord pH | 5 minutes
Small for gestational age (SGA) | 5 minutes
  it refers to an estimated fetal weight of less than the 10th percentile
Large for gestational age (LGA) | 5 minutes
  it refers to an estimated fetal weight of more than the 95th percentile

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Jani, MD, Principal Investigator — CHU Brugmann
Locations (4):
- CHU Brugmann, Brussels, Belgium
- France (2):
  - Antoine Béclère Hospital, Clamart
  - Hôpital Louis Mourier, Colombes
- Fondazione Policlinico Universitario Agostino Gemelli, Roma, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Badr DA, Mattern J, Carlin A, Cordier AG, Maillart E, El Hachem L, El Kenz H, Andronikof M, De Bels D, Damoisel C, Preseau T, Vignes D, Cannie MM, Vauloup-Fellous C, Fils JF, Benachi A, Jani JC, Vivanti AJ. Are clinical outcomes worse for pregnant women at >/=20 weeks' gestation infected with coronavirus disease 2019? A multicenter case-control study with propensity score matching. Am J Obstet Gynecol. 2020 Nov;223(5):764-768. doi: 10.1016/j.ajog.2020.07.045. Epub 2020 Jul 27. No abstract available. PMID 32730899
- [Background] Allotey J, Stallings E, Bonet M, Yap M, Chatterjee S, Kew T, Debenham L, Llavall AC, Dixit A, Zhou D, Balaji R, Lee SI, Qiu X, Yuan M, Coomar D, Sheikh J, Lawson H, Ansari K, van Wely M, van Leeuwen E, Kostova E, Kunst H, Khalil A, Tiberi S, Brizuela V, Broutet N, Kara E, Kim CR, Thorson A, Oladapo OT, Mofenson L, Zamora J, Thangaratinam S; for PregCOV-19 Living Systematic Review Consortium. Clinical manifestations, risk factors, and maternal and perinatal outcomes of coronavirus disease 2019 in pregnancy: living systematic review and meta-analysis. BMJ. 2020 Sep 1;370:m3320. doi: 10.1136/bmj.m3320. PMID 32873575
- [Background] Khalil A, von Dadelszen P, Draycott T, Ugwumadu A, O'Brien P, Magee L. Change in the Incidence of Stillbirth and Preterm Delivery During the COVID-19 Pandemic. JAMA. 2020 Jul 10;324(7):705-6. doi: 10.1001/jama.2020.12746. Online ahead of print. PMID 32648892
- [Background] Prabhu M, Cagino K, Matthews KC, Friedlander RL, Glynn SM, Kubiak JM, Yang YJ, Zhao Z, Baergen RN, DiPace JI, Razavi AS, Skupski DW, Snyder JR, Singh HK, Kalish RB, Oxford CM, Riley LE. Pregnancy and postpartum outcomes in a universally tested population for SARS-CoV-2 in New York City: a prospective cohort study. BJOG. 2020 Nov;127(12):1548-1556. doi: 10.1111/1471-0528.16403. Epub 2020 Aug 13. PMID 32633022
- [Background] Berghella V, Boelig R, Roman A, Burd J, Anderson K. Decreased incidence of preterm birth during coronavirus disease 2019 pandemic. Am J Obstet Gynecol MFM. 2020 Nov;2(4):100258. doi: 10.1016/j.ajogmf.2020.100258. Epub 2020 Oct 15. No abstract available. PMID 33083779
- [Background] Mendoza M, Garcia-Ruiz I, Maiz N, Rodo C, Garcia-Manau P, Serrano B, Lopez-Martinez RM, Balcells J, Fernandez-Hidalgo N, Carreras E, Suy A. Pre-eclampsia-like syndrome induced by severe COVID-19: a prospective observational study. BJOG. 2020 Oct;127(11):1374-1380. doi: 10.1111/1471-0528.16339. Epub 2020 Jun 21. PMID 32479682
- [Background] Cosma S, Carosso AR, Cusato J, Borella F, Carosso M, Bovetti M, Filippini C, D'Avolio A, Ghisetti V, Di Perri G, Benedetto C. Coronavirus disease 2019 and first-trimester spontaneous abortion: a case-control study of 225 pregnant patients. Am J Obstet Gynecol. 2021 Apr;224(4):391.e1-391.e7. doi: 10.1016/j.ajog.2020.10.005. Epub 2020 Oct 8. PMID 33039396